CLINICAL TRIAL: NCT02208648
Title: Coronary Assessment for Mortality Prediction
Acronym: CAMP
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/P/108
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Peri-operative Mortality; Coronary Artery Calcium
Keywords: coronary calcification; Computed Tomography; Coronary artery calcium; calcium scores; post-operative mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Deceased: Peri-operative mortality (within 90 days). Pairs of CT scans (deceased plus matched control) will be anonymised and stored on a secure server. Abbreviated Calcium scores will be generated for all patients in the trial by a trained radiologist using a calcium scoring method. The radiologist will be blinded to the group that the patient belongs to, to minimise bias. Scans (deceased patients and matched controls) will be analysed in batches of 30 pairs. Radiologist (s) will be blinded to group allocation. Scans will not be "paired" at the time of reading.
- Matched control: Patients who survived beyond 90 days peri-operatively. Pairs of CT scans (deceased plus matched control) will be anonymised and stored on a secure server. Abbreviated Calcium scores will be generated for all patients in the trial by a trained radiologist using a calcium scoring method. The radiologist will be blinded to the group that the patient belongs to, to minimise bias. Scans (deceased patients and matched controls) will be analysed in batches of 30 pairs. Radiologist (s) will be blinded to group allocation. Scans will not be "paired" at the time of reading.

SUMMARY:
The study will investigate whether the presence of coronary artery calcium as demonstrated on pre-operative, thoracic staging Computed Tomography (CT) is an independent risk factor for 90 day mortality in patients undergoing major abdominal surgery.

The study research question: Do higher levels of coronary calcification correlate to an increased risk of post-operative mortality in patients undergoing major abdominal surgery?

DETAILED DESCRIPTION:
The study uses a retrospective observational study design.

Due to the nature of the subject of the study and its retrospective design no patient contact will be necessary and all imaging reviewed will have been acquired as part of their routine level of care.

Plan for the gathering of study data

A list of patients with the following surgical codes will be identified from the hospital surgical performance database to create retrospective dataset of 5 years' worth of cases (to December 2013). This date range may be extended to ensure an adequate sample size. :

Surgical codes (Healthcare Resource Groups (HRG) codes) to be included:

F31 Large Intestine - Complex Procedures F32 Large Intestine - Very Major Procedures F33 Large Intestine - Major Procedures with complications and comorbidities (w cc) F34 Large Intestine - Major Procedures without complications and comorbidities (w/o cc) F36 Large Intestinal Disorders >69 or w cc F37 Large Intestinal Disorders <70 w/o cc

F41 General Abdominal - Very Major or Major Procedures patients over 69 years of age (>69) or w cc F42 General Abdominal - Very Major or Major Procedures patients under 70 years of age (<70) w/o cc F46 General Abdominal Disorders >69 or w cc F47 General Abdominal Disorders <70 w/o cc

Cross-reference with Somerset Cancer Register and remove any who were not recognised as having bowel cancer.

This patient list will be cross-referenced with records of peri-operative mortality (within 90 days)

Propensity match each deceased patient to a patient who survived beyond 90 days. Our matching rules will be in descending order of importance :

* HRG code
* gender,
* cancer staging
* Age+/-5yrs.
* American Society of Anesthesiologists (ASA) Grade

Where there are multiple potential matches then this will be resolved by consultation between the research team members.

Pairs of CT scans (deceased plus matched control) will be procured from WebPACS (Web Picture Archival Communication System).

Scans will be anonymised and stored on a dedicated secure radiology research server.

Abbreviated Calcium scores will be generated for all patients in the trial by a trained radiologist using the calcium scoring method. Calcium burden will be recorded on a scale of 1-12 . The radiologist will be blinded to the group that the patient belongs to, to minimise bias.

Scans (deceased patients and matched controls) will be analysed in batches of 30 pairs. Radiologist (s) will be blinded to group allocation. Scans will not be "paired" at the time of reading.

Interim statistical analysis (of calcium scores) will be performed after each batch of scans.

ELIGIBILITY:
Inclusion Criteria:

* All adults ≥18yrs old
* Major abdominal surgery (See HRG Codes)
* Bowel Cancer
* Elective admission

Exclusion Criteria:

* <18 yrs old
* No suitable matched patient
* No CT Chest available
* Emergency admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Plymouth Hospital NHS Trust patients
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is an abbreviated calcium score | 5 years
  To investigate whether the presence and severity of coronary calcification identified on routine, pre-operative staging CT scans of the chest are an independent risk factor for patients undergoing major surgery. Techniques have now been validated where calcium scores can be estimated from routine CT scans of the chest (Shemesh et al. 2006).

SECONDARY OUTCOMES:
To assess the use of the calcium scoring technique in contrast enhanced studies. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl Roobottom, MBChB(Hons), Study Chair — Plymouth Hospital NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

REFERENCES:
- [Background] Shemesh J, Henschke CI, Farooqi A, Yip R, Yankelevitz DF, Shaham D, Miettinen OS. Frequency of coronary artery calcification on low-dose computed tomography screening for lung cancer. Clin Imaging. 2006 May-Jun;30(3):181-5. doi: 10.1016/j.clinimag.2005.11.002. PMID 16632153